CLINICAL TRIAL: NCT01351740
Title: Switch to Unboosted Atazanavir With Tenofovir (SUAT) Study
Brief Title: Switch to Unboosted Atazanavir With Tenofovir Study
Acronym: SUAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Marianne Harris, MD, Dr. Marianne Harris, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H10-03255; H10-03255 (Other: UBC/Providence Health Care REB)
Record Dates: First submitted 2011-05-09; First posted 2011-05-11 (Estimated); Results first posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2017-10

CONDITIONS: HIV Infection
Keywords: HIV; Anti-HIV Agents; HIV Protease Inhibitors
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate; atazanavir, ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Switch (Experimental): switch to unboosted atazanavir 400mg daily with the same nucleoside (NRTI) backbone
  Interventions: Drug: atazanavir
- Continuation (Active Comparator): continue on current regimen of atazanavir/ritonavir 300mg/100mg with the same nucleoside (NRTI) backbone
  Interventions: Drug: atazanavir/ritonavir

INTERVENTIONS:
Drug: atazanavir — switch to unboosted atazanavir 400 mg daily
  Arms: Switch
Drug: atazanavir/ritonavir — Continue current regimen of atazanavir 300 mg/ ritonavir 100 mg daily
  Arms: Continuation

SUMMARY:
A drug-drug interaction between the anti-HIV drugs tenofovir DF (TDF) and atazanavir (ATZ) results in lower ATZ plasma levels when the drugs are given together, particularly in patients not taking ritonavir to boost ATZ levels. Lower plasma drug levels may make the anti-HIV regimen less effective in controlling the HIV virus levels in the blood. For this reason, current treatment guidelines recommend that ATZ always be boosted with ritonavir in regimens also containing TDF. However, withdrawal of ritonavir is often desirable given the tolerability and toxicity issues with this agent, even at the low dose (100 mg daily) used to boost ATZ. For example, ritonavir can cause stomach upset, nausea, diarrhea, high cholesterol levels, and liver enzyme abnormalities.

However, there is evidence that plasma ATZ levels may not predict treatment success on unboosted ATZ regimens, particularly among people whose plasma HIV virus is already under control and unboosted ATZ is being used as a maintenance strategy. In the BC Centre for Excellence in HIV/AIDS Drug Treatment Program (DTP), nearly 100 patients originally treated with ritonavir-boosted ATZ + TDF (+ FTC or 3TC) are receiving successful maintenance therapy with unboosted ATZ and the same TDF-based backbone.

The study will examine the hypothesis that switching to maintenance therapy with unboosted ATZ 400mg daily will have similar 48-week virologic efficacy to continuing ATZ/ritonavir 300/100mg daily among HIV-infected adults with stable viral load suppression on regimens comprising ATZ/ritonavir 300/100mg daily with TDF plus either FTC or 3TC, despite potentially lower ATZ trough levels with the unboosted regimen. In other words, patients whose HIV viral load is undetectable while receiving TDF (+FTC or 3TC) and ATZ/ritonavir will continue to maintain an undetectable viral load after switching to unboosted ATZ without ritonavir, in the same proportions as those continuing on their boosted ATZ/ritonavir regimen.

DETAILED DESCRIPTION:
Following a screening visit to establish study eligibility, eligible consenting subjects will be randomized 1:1 to one of the two treatment arms (switch to unboosted ATZ or continue ritonavir-boosted ATZ). Randomized open-label treatment will commence following study procedures at baseline. Participants will be assessed at baseline and at weeks 4, 8, 12, 24, 36, and 48. On-study evaluations will include assessment of adverse clinical events and medication changes; blood tests for HIV viral load, CD4 cell count, standard safety parameters, fasting lipids and glucose, and pregnancy testing (if applicable); and urine tests for urinalysis and albumin to creatinine ratio. In addition, a serum sample will be stored at each visit for possible future testing. A timed plasma sample for measurement of pre-dose trough ATZ levels will be obtained once per subject at 4-8 weeks. Quality of life will be assessed by completion of the MOS-HIV questionnaire at baseline and every 12 weeks. Adherence will be assessed based on prescription refill data.

In case of protocol-defined virologic failure, a plasma sample for ATZ trough level will be collected, and genotypic resistance testing will be performed on plasma samples with viral load >250 copies/mL. Subjects with confirmed virologic failure will be asked to come to the clinic and will have their HIV treatment changed to a more effective regimen, selected based on the results of genotypic testing, as soon as possible.

The anticipated rate of confirmed virologic failure in the control arm is no more than 15% over the 48 weeks of the study. Once at least 20 subjects have been assigned to the experimental (switch) treatment arm, if the observed confirmed virologic failure rate in the experimental arm is greater than twice this rate, i.e. >30%, at any time during the study, the study will be stopped. At this time, subjects in the experimental arm will be reassessed as soon as possible and will resume ritonavir-boosted atazanavir or other effective HIV therapy as appropriate. The failure rate will be reassessed at a minimum after each 20 subjects are enrolled into the experimental (switch) arm.

ELIGIBILITY:
Inclusion Criteria:

1. HIV infected adults at least 19 years of age
2. Willing and able to provide informed consent to study participation
3. Currently receiving a regimen including atazanavir 300mg/ritonavir 100mg daily with either tenofovir/emtricitabine (FTC) or tenofovir/lamivudine (3TC), for at least 3 months
4. Plasma viral load (VL) <40 copies/mL for at least 2 consecutive measurements including the screening value, and < 150 copies/mL continuously for at least 3 months prior to screening
5. Current regimen is first antiretroviral regimen, or if not first regimen, no evidence of resistance to any nucleosides (NRTIs) or protease inhibitors (PIs) on previous resistance tests
6. Any CD4

Exclusion Criteria:

1. Clinically significant intolerance or toxicity with current regimen precluding regimen continuation (e.g. intolerance/toxicity to ritonavir necessitating ritonavir discontinuation)
2. pregnancy or breast-feeding
3. antiretroviral regimen including any nonnucleoside reverse transcriptase inhibitor (nevirapine, efavirenz, or etravirine)
4. antiretroviral regimen including any protease inhibitor other than atazanavir and ritonavir
5. concomitant treatment with proton pump inhibitors, rifampin, St. John's wort, or garlic supplements. (Antacids and H2 receptor antagonists will be allowed provided their dosing is separated from atazanavir administration by at least 2 and 10 hours, respectively).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-07; Primary Completion 2015-01 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Harris, MD, Principal Investigator — Providence Health Care/ University of British Columbia
Locations (1):
- Immunodeficiency Clinic, St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Result] Harris M, Ganase B, Watson B, Hull MW, Guillemi SA, Zhang W, Saeedi R, Harrigan PR. Efficacy and safety of "unboosting" atazanavir in a randomized controlled trial among HIV-infected patients receiving tenofovir DF. HIV Clin Trials. 2017 Jan;18(1):39-47. doi: 10.1080/15284336.2016.1271503. Epub 2017 Jan 9. PMID 28067119

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Switch | Continuation
Started | 25 | 25
Completed | 23 | 19
Not Completed | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Switch: Switch to atazanavir 400 mg daily
- Continuation: Remain on atazanavir/ritonavir 300mg/100 mg daily
- Total: Total of all reporting groups
Arm/Group | Switch | Continuation | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 48 [42 to 52] | 46 [39 to 53] | 47 [40 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Proportions of Subjects Experiencing Virologic Failure by Randomized Treatment Arm
Description: For the purposes of the study, virologic failure is defined as either regimen change for any reason, or plasma viral load >400 copies/mL on 2 consecutive measurements >2 weeks apart.
Time Frame: at or before 48 weeks.
Measure: Count of Participants; unit: Participants
Groups:
- Continuation: Remain on atazanavir/ritonavir 300mg/100mg daily
Arm/Group | Switch | Continuation
Number analyzed (Participants) | 25 | 25
Participants | 2 | 6

2. Secondary Outcome: Proportions of Subjects in Each Randomized Treatment Arm With Atazanavir Trough Levels Below 150ng/mL
Description: Therapeutic drug monitoring (TDM) to determine atazanavir trough plasma level will be performed once on all subjects at 4-8 weeks
Time Frame: 1 month (4-8 weeks)
Measure: Count of Participants; unit: Participants
Groups:
- Continuation: Remain on atazanavir/ritonavir 300mg/100mg
Arm/Group | Switch | Continuation
Number analyzed (Participants) | 24 | 12
Participants | 14 | 3

3. Secondary Outcome: Proportion of Subjects Experiencing Virologic Failure by Results of 1-month TDM
Description: For the purposes of the study, virologic failure is defined as either regimen change for any reason, or plasma viral load >400 copies/mL on 2 consecutive measurements >2 weeks apart. Comparison will be made between subjects with 1-month (4-8 week) on-study atazanavir trough levels <150ng/mL and those with 1-month (4-8 week) on-study atazanavir trough levels >150ng/mL.
Time Frame: at or before 48 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Proportions of Subjects Experiencing Virologic Failure by Randomized Treatment Arm
Description: as for outcome 1
Time Frame: at or before 24 weeks.
Reporting Status: Not Posted

5. Secondary Outcome: Proportion of Subjects Experiencing Virologic Failure by Results of 1-month TDM
Description: as for outcome 3
Time Frame: at or before 24 weeks
Reporting Status: Not Posted

6. Secondary Outcome: CD4 Cell Count Changes (Absolute and Fraction)
Description: Comparison will be made between randomized treatment arms.
Time Frame: 24 and 48 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Safety (Clinical and Laboratory Adverse Events)
Description: Serious adverse events and discontinuations will be compared between randomized treatment arms
Time Frame: 24 and 48 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Total Serum Bilirubin Levels
Description: Comparison will be made between randomized treatment arms.
Time Frame: 24 and 48 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Metabolic Parameters
Description: Comparison will be made between randomized treatment arms with respect to changes in fasting lipids and glucose, highly sensitive C-reactive protein [hsCRP], and apolipoprotein [apo]B, and proportions of subjects developing abnormalities or crossing predefined limits (e.g. NCEP thresholds for lipids)
Time Frame: 24 and 48 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Quality of Life as Assessed by MOS-HIV
Description: Changes in MOS-HIV scores from baseline will be compared between randomized treatment arms.
Time Frame: 24 and 48 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 48 weeks
Groups:
- Continuation: Remain on atazanavir/ritonavir 300 mg/100 mg daily
Arm/Group | Switch | Continuation
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 3/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Switch (N=25) | Continuation (N=25)
diarrhea (Gastrointestinal disorders) | 0 | 1
renal toxicity (Renal and urinary disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes